CLINICAL TRIAL: NCT03722615
Title: Epidemiology of Congenital Cytomegalovirus in a High HIV Prevalence Setting, South Africa
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Jayani Pathirana, PhD Fellow, University of Witwatersrand, South Africa
Other Study IDs: M151161
Record Dates: First submitted 2018-10-19; First posted 2018-10-29 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Cytomegalovirus Congenital; Hearing Loss; Neurodevelopmental Disorders; Immunogenicity; Neonatal Death; Stillbirth
MeSH Terms: conditions — Cytomegalovirus Infections; Hearing Loss; Neurodevelopmental Disorders; Perinatal Death; Stillbirth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this project is to determine the epidemiology of congenital cytomegalovirus (CMV) infection and incidence of subsequent permanent neurological sequelae in a high HIV prevalent setting in Soweto, Johannesburg. A cross-sectional study will be conducted on mother-infant pairs, screening mothers for CMV infection and newborns for congenital CMV infection. Maternal CMV prevalence will be determined by testing for CMV specific antibodies in blood. Newborn congenital infection will be determined by polymerase chain reaction (PCR) tests on newborn saliva and urine within 3 weeks of birth. Various risk factors associated with congenital CMV such as HIV exposure, and gestational age will be assessed. The association between maternal vaginal CMV shedding postnatally with congenital CMV infection will be explored by swabbing maternal vaginal fluid and conducting quantitative CMV PCR analysis. Newborns confirmed with congenital CMV and a control group of uninfected newborns will form a cohort to be followed up until 12 months of age monitoring for various neurological sequelae such as hearing loss, neurodevelopmental impairment, ocular damage, cerebral damage and seizures.

A comparison of vaccine immune responses between cases of congenital CMV and the CMV uninfected infants to the primary series of vaccines in the National Expanded Programme on Immunisation will be compared. The contribution of CMV infection to neonatal death and stillbirths will be described by minimally invasive tissue sampling (MITS) for CMV on babies that die during the neonatal period and stillbirths.

ELIGIBILITY:
Inclusion Criteria:

* Mother's age ≥18y
* Residing in Soweto and would be available for study follow-up
* Consents to enrol self and baby in study

Exclusion Criteria:

- Mother not enrolled in V98_28OBTP (NCT02215226)

Ages: 1 Minute to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns of women aged 18 years or older born at Chris Hani Baragwanath Academic hospital in the Johannesburg area enrolled in V98_28OBTP (NCT02215226).
  Stillbirths and Neonatal deaths at Chris Hani Baragwanath Academic hospital in the Johannesburg area.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of congenital cytomegalovirus infection in HIV exposed and HIV unexposed newborns | May 2016 - December 2016
  Prevalence will be determined by testing a saliva sample collected at birth for CMV DNA by polymerase chain reaction (PCR) assay. Newborns that test positive for CMV at birth will have confirmatory testing done within 3 weeks of birth by testing a repeat saliva and urine sample for CMV DNA by PCR. Confirmed cases will be divided by the total number of newborns screened, stratified by HIV exposure status to determine CMV prevalence.
Incidence of sensorineural hearing loss in congenital CMV infected and uninfected infants, assessed by visual reinforced audiometry | May 2016 - May 2019
  Screening for sensorineural hearing loss is initially conducted by acoustic reflex testing (ART) and distortion product otoacoustic emissions (DPOAE). To pass ART testing, the infant will have to obtain at least two reflexes at either 0.5, 1, 2 and/or 4kHz in both ears. To pass DPOAE testing, the infant will have to pass at least 3 frequencies (2,3,4 and/or 5kHz) in both ears, which is an overall pass. If any of ART or DPOAE has not been passed, the child will have diagnostic visual reinforced audiometry. Hearing thresholds will be defined as: 0 to 20 dB for normal hearing, 21 to 45 dB for mild hearing loss, 46 to 70 dB for moderate hearing loss, and 71 dB or higher for severe hearing loss.
Incidence of neurodevelopmental delay in congenital CMV infected and uninfected children at one year of age assessed by scores obtained in the Bayley III developmental assessment tool. | May 2017 to March 2018
  The Bayley III scales of infant and toddler development assess the neurodevelopmental domains based on observed responses to a set of tasks presented to the child which are scored directly on the following subscales: cognitive scale, language summed scale of receptive and expressive language subscales and motor summed scale of fine and gross-motor subscales. Composite scores are derived from raw scores for cognitive, language, and motor development and scaled to a metric, with a mean of 100, standard deviation of 15, and range of 40 to 160. Performance that is 2.0 or more standard deviations below the mean score for each group will be used to define neurodevelopmental delay at 6 and 12 months.

SECONDARY OUTCOMES:
Prevalence of CMV infection in stillbirths and neonatal deaths | July 2015 to August 2016
  Prevalence of in-utero CMV infection in stillbirths and neonatal deaths (occurring before 3 weeks age) and sites of infection. Minimally invasive tissue sampling of the major organs (lungs, brain, liver) and cerebrospinal fluid and blood samples will be tested for CMV by PCR assay.
Immunogenicity to primary series of childhood vaccinations in congenital CMV infected and uninfected children | October 2016 to February 2018
  When infants are aged 6 months a venous blood sample will be collected. Antibody to diphtheria toxoid, tetanus-toxoid, pertussis toxoid, filamentous hemagglutinin (FHA) and hepatitis B surface antigen (HBsAg) will be measured by an in-house Luminex multiplex immunoassay. Immune responses to the primary series of PCV will be measured by a standardized enzyme immunoassay (EIA) to test for vaccine serotype-specific capsular immunoglobulin (Ig) G antibody concentrations and opsonophagocytic assay.

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, Study Director — Univeristy of Witwatersrand, South Africa
Locations (1):
- Respiratory and Meningeal Pathogen Research Unit, Soweto, Johannesburg, South Africa

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT03722615/Prot_SAP_000.pdf